CLINICAL TRIAL: NCT04430231
Title: Does Delaying Curative Surgery for Colorectal Cancer Influence Long-term Disease Free Survival.: A COHORT STUDY
Brief Title: Does Delaying Curative Surgery for Colorectal Cancer Influence Long-term Disease Free Survival.
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Stephanie Garcia Botello, Clinical Professor, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: 2019/285
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Wait list time 0-2 weeks: Wait list time 0-2 weeks
  Interventions: Other: Wait list time
- Wait list time 2-4 weeks: Wait list time 2-4 weeks
  Interventions: Other: Wait list time
- Wait list time 4-6 weeks: Wait list time 4-6 weeks
  Interventions: Other: Wait list time
- Wait list time > 6 weeks: Wait list time > 6 weeks
  Interventions: Other: Wait list time

INTERVENTIONS:
Other: Wait list time

SUMMARY:
This work is an original clinical research article describing the relationship between wait list tome for colorectal cancer patients and long-term survival. These findings are particularly relevant for management of surgical wait lists during crisis such as the Covid-19 pandemic. The lack of a relationship between wait list time and disease free survival and tendency for improved survival in the 4-6 week imply some colorectal cancer operations can be safely delayed during times of limited resources.

DETAILED DESCRIPTION:
Background Surgical wait list time is a major problem in many health-care systems and its influence on survival is unclear. The aim of this study is to assess the impact of the wait list time on long term disease-free survival in patients scheduled for colorectal cancer resection.

Materials and Methods A prospective, single center study was carried out in patients with stage I-III colorectal cancer scheduled for surgery between 2012-2017 at a Colorectal Surgery Unit of a tertiary care center. Wait list time was defined as the time from completion of diagnostic workup and definitive surgery and divided into 2-week intervals from 2 to 6 weeks. The outcome variables were 2- and 5-year disease free survival. Screening for disease progression was with carcinoembryonic antigen levels and chest/abdominal computed tomography scan. Data was collected prospectively and subsequently analyzed.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) stage I through III confirmed adenocarcinomas
* With "colon" or "upper rectum" as their primary site of malignancy according to International Classification of Diseases for Oncology, Third Edition topography code.

Exclusion Criteria:

* Emergency surgery,
* More than one primary site,
* Synchronous metastasis or peritoneal carcinomatosis at the time of surgery
* If they received neoadjuvant chemoradiotherapy
* If they had a local transanal excision.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had American Joint Committee on Cancer (AJCC) stage I through III confirmed adenocarcinomas were selected, with "colon" or "upper rectum" as their primary site of malignancy according to International Classification of Diseases for Oncology, Third Edition topography code.
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Disease-free overall survival | 5 years

IPD SHARING:
Plan to Share IPD: Undecided